CLINICAL TRIAL: NCT01744756
Title: Interventional Trial of Subconjunctival Bevacizumab in Recurrent Pterygium
Brief Title: Subconjunctival Bevacizumab and Recurrent Pterygium
Acronym: BRP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pterygium bevacizumab
Record Dates: First submitted 2012-11-29; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Pterygium
Keywords: Subconjunctival Bevacizumab; Recurrent pterygium
MeSH Terms: conditions — Pterygium | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subconjunctival Bevacizumab (Experimental): One aplication of subconjunctival Bevacizumab 0,5 ml
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — One subconjunctival aplication of Bevacizumabe 0,5ml
  Other Names: Avastin

SUMMARY:
A study to research whether subconjunctival bevacizumab injection may potentially suppress neovascularization in pterygium, retarding and decreasing the size of recurrent pterygium.

DETAILED DESCRIPTION:
1. Pacients with recurrent pterygium
2. Anti-VEGF therapy -Bevacizumab

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pterygium

Exclusion Criteria:

* Pregnant or lactating women
* History of myocardial infarction
* History of stroke

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pterygium size after subconjunctival bevacizumab | 8 weeks
  -Size of recurrent pterygium (measured in mm) after injection

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  -Number of patients with hyposphagma and irritative symptoms after subconjunctival injection

CONTACTS AND LOCATIONS:
Overall Officials: Larissa S Stival, MD, Study Chair — Instituto de Olhos de Goiania
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil

REFERENCES:
- [Derived] Stival LR, Lago AM, Figueiredo MN, Bittar RH, Machado ML, Nassaralla Junior JJ. Efficacy and safety of subconjunctival bevacizumab for recurrent pterygium. Arq Bras Oftalmol. 2014 Jan-Feb;77(1):4-7. doi: 10.5935/0004-2749.20140003. PMID 25076364